CLINICAL TRIAL: NCT03025971
Title: Efficacy and Safety Evaluation for The Interventional Aortic Valve Bioprosthesis and Delivery System in Patients With Severe Aortic Stenosis and/or Aortic Regurgitation With Elevated Surgical Risk
Brief Title: Safety & Efficacy of the J-Valve Ausper System in Patients With Severe Aortic Stenosis and/or Aortic Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JC Medical, Inc., an affiliate of Edwards Lifesciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S20131216
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Disease
Keywords: Severe Aortic Stenosis and/or severe aortic regurgitation
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm observational study (Other): Intervention: J-Valve Transcatheter Aortic valve replacement. Prospective, multi-center, single arm observational study. Subjects will include patients with severe aortic valve stenosis and/or severe aortic regurgitation who require replacement of their native aortic valve.
  Interventions: Device: J-Valve Transcatheter Aortic valve replacement

INTERVENTIONS:
Device: J-Valve Transcatheter Aortic valve replacement — Transapical Transcatheter Aortic Valve Replacement
  Other Names: TAVI

SUMMARY:
A prospective, multicenter, nonrandomized, single-arm, clinical study.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the J-Valve Ausper system for the treatment of patients with severe aortic stenosis and/or aortic regurgitation with elevated risk for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Age ≥18years of age
3. Presents with symptomatic aortic stenosis and/or aortic regurgitation, as well as NYHA rating of NYHA ≥ II
4. Has undergone the diagnosis of at least one interventional cardiologist and two cardiac surgeons: the patients are contraindicated for traditional open heart valve replacement surgery (defined as 30 days post-op mortality risk >50%, irreversible complications, or other influential post-operative factors [such as severe calcification in the ascending aorta and aortic valve, weak physical condition, chest deformities, severe liver diseases, severe lung diseases, etc.] or high risk for surgery (LogEuroSCORE≥20% and or STS≥8)
5. Has a diagnosis from at least one interventional cardiologist and two cardiac surgeons that the patient may benefit from a valve implantation
6. Severe aortic stenosis with electrocardiography results as follows: mean transvalvular pressure gradient ≥40 mmHg or maximal forward aortic blood flow velocity of ≥4.0 m/s, aortic valve area < 0.8 cm2 (or AVA index < 0.5 cm2/m2); and/or severe aortic regurgitation, electrocardiography results show symptomatic moderate regurgitation or severe regurgitation
7. Without severe pulmonary arterial hypertension
8. The patient is willing to cooperate with all follow-up visits.

   Anatomical Inclusion Criteria:
9. Aortic annulus >19mm and <29mm, standardized using cardiac CT measurements;
10. Ascending aortic diameter <50mm at the sinotubular junction.

Exclusion Criteria:

1. Patients with infection or who have any sign of infection
2. Previous history of endocarditis or patients with active endocarditis
3. Incidence of acute myocardial infarction within the past 30 days (Q-wave MI, or non Q-wave MI with creatine kinase, an increase in troponin T)
4. Any cardiac mass discovered during echocardiography, left ventricular or atrial thrombosis
5. Suffering from uncontrollable atrial fibrillation
6. Hereditary hypertrophic cardiomyopathy
7. Mitral or tricuspid valve insufficiency (Class Ⅱ regurgitation or greater)
8. Has previously undergone aortic valve implantation (mechanical valve or biological valve frame)
9. Is known to be allergic to contrast agents, aspirin, heparin, ticlopidine medications, nitinol or porcine products
10. Is known to be contraindicated for or is allergic to all anti-coagulants or is unable to use anti-coagulants during the study
11. Is known to have one of the following conditions (according to evaluations beginning from screening through the day of the procedure):

    * Other diseases that may reduce the life expectancy to less than 12 months (such as clinically recurrent or metastatic cancer, congestive heart failure, etc.)
    * Currently has drug abuse problems (such as alcohol, cocaine, heroin, etc.)
    * Plans to undergo surgery that may result in non-compliance with the study protocol or that may cause confusion in data interpretation.
12. Has experienced a cerebrovascular accident (CVA) within the last 6 months
13. Patients suffering from stenosis of the carotid, internal carotid, or vertebral arteries (70%)
14. White cell count <3×109/L, platelet count<50×109/L
15. Hemoglobin <90 g/L
16. Severely lowered left ventricular function, left ventricular ejection fraction < 20 %
17. Aortic aneurysm in the abdomen or chest
18. Hepatic encephalopathy or acute active hepatitis
19. Currently undergoing dialysis or baseline creatine levels >2.5 mg/dL (221μmoI/L)
20. Prone to bleeding, has a history of clotting disorders or refuses blood transfusions
21. Active ulcer or active gastrointestinal (GI) bleeding
22. Suffering from nervous system diseases that severely influence the patients' ability to move or to perform daily activities
23. Patients with severe dementia
24. Any reason for emergent surgery
25. Taking part in other clinical trials for pharmaceuticals or medical devices
26. Those who are pregnant, plan to become pregnant, or who are taking estrogen or estrogen-like drugs (women suspected of being pregnant must test negative on a urine pregnancy test or for chorionic gonadotropin serum).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality | 12 months

SECONDARY OUTCOMES:
Cardiac function improvement | 30 days, 6 months, 12 months and annually up to 5 years
  New York Heart Association (NYHA) Functional class

OTHER OUTCOMES:
Incidence of Major Adverse Cardiovascular Cerebrovascular Events (MACCE) | 30 days, 6 months, 12 months and annually up to 5 years
  All-cause mortality, myocardial infarction (Q-wave and non Q-wave), stroke, acute renal damage, major vascular complications, life-threatening bleeding events, or re-operation due to valvular dysfunction (surgical or interventional treatment).
Incidence of Major Adverse Valve Related Events (MAVRE) | 30 days, 6 months, 12 months and annually up to 5 years
  Valve related deaths, valve related complications, or implantation of a permanent pacemaker or defibrillator within 14 days of operation. Valve related complications include any structural degradation or non-structural dysfunction of the valve prosthesis, thrombosis, embolism, bleeding events, or valve prosthesis endocarditis.
Technical Success | Within 30 days post procedure
  * Implantation of the valve into the precise anatomical position of the native aortic valve.
  * No valve migration
  * No positioning errors.
  * Paravalvular leak is less than moderate (ratio of regurgitation surface area/left ventricular surface area 25-50%).
  * Successful removal of the entire delivery device.
  * Implantation of the valve into the precise anatomical position of the native aortic valve.
  * No valve migration
  * No positioning errors.
  * Paravalvular leak is less than moderate (ratio of regurgitation surface area/left ventricular surface area 25-50%).
  * Successful removal of the entire delivery device.
Device Success | Within 30 days post procedure
  * no intraoperative death,
  * valve prosthesis has been accurately implanted into the anatomic position of the native aortic valve is performing its anticipated function.
  * The intended performance of the bioprosthetic valve function:
    * no mismatch between the valve prosthesis and the patient,
    * mean transvalvular pressure gradient is ≤20 mmHg or
    * peak forward aortic blood flow velocity of <3.0 m/s, and no moderate or severe aortic regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhang, MD, Study Director — CEO, President
Locations (3):
- China (3):
  - West China Hospital, Chengdu
  - Zhongshan Hospital, Shanghai
  - Fuwai Cardiovascular Hospital, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided